CLINICAL TRIAL: NCT04593550
Title: A Pilot Study to Identify Electroencephalographic Changes Under General Anesthesia in Patients With and Without History of Chemotherapy
Brief Title: Electroencephalographic Changes Under General Anesthesia in Patients With Gynecologic Cancers With and Without History of Chemotherapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1120; NCI-2020-06076 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1120 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-29; First posted 2020-10-20 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (BrainCheck, 3D-CAM, EEG): Patients undergo cognitive function assessment BrainCheck over 10 minutes before surgery, day 1 after surgery, and day 2 after surgery (if patients are still admitted to the hospital) and 3D-confusion assessment over 10 minutes BID on day 1 after surgery and day 2 after surgery (if patients are still admitted to the hospital). Patients also undergo EEG during surgery and collection of blood samples 30-60 minutes after surgery.
  Interventions: Procedure: Biospecimen Collection; Behavioral: BrainCheck Cognitive Assessment; Procedure: Cognitive Assessment; Procedure: Electroencephalography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Behavioral: BrainCheck Cognitive Assessment — Undergo cognitive function assessment BrainCheck
  Other Names: BrainCheck
Procedure: Cognitive Assessment — Undergo 3D-Confusion assessment
Procedure: Electroencephalography — Undergo EEG
  Other Names: EEG; electroencephalogram

SUMMARY:
This study compares changes in brain waves in women with gynecologic cancers who have or have not received chemotherapy and who are scheduled to receive surgery as part of their standard care. Electroencephalography is a test that measures brain waves and may help learn if sensitivity to anesthesia is higher in women who have received chemotherapy than women who have not. This study may help researchers learn if receiving chemotherapy before surgery can affect the way the brain responds to anesthesia during and after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess electroencephalography (EEG) changes of women with and without history of chemotherapy exposure undergoing volatile general anesthesia.

SECONDARY OBJECTIVE:

I. To evaluate if chemotherapy-induced cognitive impairment is associated with an increased sensitivity to general anesthetic agents captured by the patient state index (PSI) and observable in changes in alpha (8-12 H) activity in the frontal regions of the EEG) and other study features such as EEG power, burst suppression analysis, burst suppression ratio, and coherence analysis.

EXPLORATORY OBJECTIVES:

I. To assess the relationship between preoperative cognitive function and electroencephalographic changes under general anesthesia.

II. To assess the relationship between EEG signatures under general anesthesia and postoperative cognitive function.

III. To collect blood specimens for extracting information on serum lipids and cytokines at two different times, before anesthetic induction, and 30 to 60 minutes upon arrival to the postoperative anesthesia care unit.

OUTLINE:

Patients undergo cognitive function assessment BrainCheck over 10 minutes before surgery, day 1 after surgery, and day 2 after surgery (if patients are still admitted to the hospital) and 3D-confusion assessment over 10 minutes twice daily (BID) on day 1 after surgery and day 2 after surgery (if patients are still admitted to the hospital). Patients also undergo EEG during surgery and collection of blood samples 30-60 minutes after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Women between 40-60 years of age; with or without history of systemic chemotherapy;
3. American Society of Anesthesiologists physical status (ASA) 1-3;
4. Scheduled surgery: open gynecologic surgery;
5. Able to complete all study questionnaires.

Exclusion criteria:

1. Emergency surgery
2. ASA ≥ 4
3. Patients with extra-abdominal metastatic disease
4. Patients unable to complete preoperative and postoperative cognitive tests
5. Non-English-speaking patients

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with gynecologic cancers with or without history of preoperative chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Difference in the amplitude of alpha oscillations 15 minutes after incision | 15 minutes after incision
  Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. Will explore differences in the analysis of the alpha oscillations

SECONDARY OUTCOMES:
Patient State Index (PSI) | Up to 2 days post surgery
  For each participant, the PSI will be recorded from the SedLine monitor. Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. PSI will be analyzed between both groups of patients using an independent samples t-test or Wilcoxon's ranksum test, if more appropriate. Chi-square or Fisher's exact tests will be used if study outcomes are categorical. Finally, will also use both Pearson and Spearman's correlation to assess the association between study features such as PSI and cognitive function.
Electroencephalography (EEG) power | During surgery
  For each participant, will calculate the slow (0.1-1 Hz), delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), beta (12-25 Hz), gamma (25-40Hz), and total power (0.1-40Hz). Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. Will explore EEG power between both groups of patients using an independent samples t-test or Wilcoxon's ranksum test, if more appropriate. Chi-square or Fisher's exact tests will be used if study outcomes are categorical. Finally, will also use both Pearson and Spearman's correlation to assess the association between study features such as EEG power and cognitive function.
Burst suppression analysis | During surgery
  When delivered in a sufficiently high dose, intravenous and volatile anesthetics induce burst suppression. This will be obtained from visual inspection of EEG spectrograms. For each participant, burst suppression will be considered significant if three or more events are observed within 2 min period of stable anesthesia. Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. Will explore burst suppression between both groups of patients using an independent samples t-test or Wilcoxon's ranksum test, if more appropriate. Chi-square or Fisher's exact tests will be used if study outcomes are categorical.
Burst suppression ratio | During surgery
  Burst suppression ratio is defined as a time domain measure used to track quantitatively the level of burst suppression. It ranges from 0 to 1 and is one of the parameters used to determine depth-of- anesthesia. Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. Will explore burst suppression ratio between both groups of patients using an independent samples t-test or Wilcoxon's ranksum test, if more appropriate. Chi-square or Fisher's exact tests will be used if study outcomes are categorical. Finally, will also use both Pearson and Spearman's correlation to assess the association between study features such as burst suppression ratio for each band and cognitive function.
Coherence analysis | During surgery
  Will be calculated as a measure of synchrony between two signals at the same frequency as previously described by Purdon et al. Data will be analyzed using descriptive statistics and visualizations of the data to establish patterns of symmetry, skewness, and outliers. Will explore coherence between both groups of patients using an independent samples t-test or Wilcoxon's ranksum test, if more appropriate. Chi-square or Fisher's exact tests will be used if study outcomes are categorical.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org